CLINICAL TRIAL: NCT06786195
Title: Is the Bone Myoregulation Reflex Response to Weight-Bearing Activities Low in Senile Osteoporosis?
Brief Title: Bone Myoregulation Reflex in Senile Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Eser Kalaoglu, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IstPRMTRH-EK2
Record Dates: First submitted 2025-01-09; First posted 2025-01-22 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Osteoporosis (Senile)
Keywords: Reflex; Vibration; Bone; Loading exercise; Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: This study employs a quasi-experimental design. Diagnosis of osteoporosis was made according to the World Health Organization classification. Individuals with a T-score of -2.5 or below were classified as having osteoporosis. Participants will be divided into two groups: a group with osteoporosis (Group 1) and a group without osteoporosis (Group 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Those with osteoporosis
  Interventions: Other: Whole-body vibration and Jumping
- Group 2 (Experimental): Those without osteoporosis
  Interventions: Other: Whole-body vibration and Jumping

INTERVENTIONS:
Other: Whole-body vibration and Jumping — The subjects were first asked to jump in place 20 times, as if they were jumping rope. Then, whole-body vibration was applied. While the participants stood upright on the whole-body vibration device, low-amplitude (1.2 mm) vibrations were applied at eight different frequencies (25, 27, 29, 31, 33, 35, 37, 39 Hz), each lasting for 10 seconds, with a 5-second rest period in between. The Achilles tendon will be percussed 10 times with an electronic reflex hammer.

SUMMARY:
Osteoporosis is a systemic skeletal disease characterized by weakened and fragile bones. It often remains asymptomatic in its early stages but can lead to serious health problems, particularly fractures.The mechanostat theory explains that bone mass is regulated by mechanical loading. Increased activity stimulates bone formation, while decreased activity promotes bone resorption. The "bone reflex" concept further suggests that the nervous system plays a crucial role in this process by regulating both bone metabolism (osteoregulation) and muscle activity (myoregulation) in response to mechanical loading.

DETAILED DESCRIPTION:
Background and Objectives:Osteoporosis is a systemic skeletal disease characterized by weakened and fragile bone tissue. Typically asymptomatic in its early stages, it can lead to severe health consequences, particularly fractures. Bone mineral density (BMD) measurements, as defined by the World Health Organization, are considered the gold standard for diagnosing osteoporosis. The prevalence of osteoporosis is on the rise due to the aging population and the influence of lifestyle factors.

Recently, the bone reflex has been defined, suggesting that the central nervous system controls the local regulatory mechanisms described by Wolf and Frost. The bone reflex describes how osteocytes are stimulated by mechanical loading, leading to the neural regulation of bone formation and resorption according to mechanical needs (bone osteoregulation reflex). Additionally, it describes a mechanism by which the nervous system reflexively regulates the activity of surrounding muscles to optimally position the bone to resist applied mechanical load (bone myoregulation reflex).

Methods: This study employs a quasi-experimental design. The study will be conducted with a total of 22 patients aged 60-70, men. Diagnosis of osteoporosis was made according to the World Health Organization classification. Individuals with a T-score of -2.5 or below were classified as having osteoporosis. Participants will be divided into two groups: a group with osteoporosis (Group 1) and a group without osteoporosis (Group 2).

Procedures:

Bone myoregulation reflex activity of the soleus and tibialis anterior muscles will be assessed in both groups during whole-body vibration and jumping using surface electromyography.

* Jumping Test: Participants will be instructed to jump in place 20 times, similar to rope skipping, with a 5-second rest interval between each jump.
* Whole-Body Vibration: Participants will stand on the plate and undergo low-amplitude (1.2 mm) whole-body vibration at eight different frequencies (25, 27, 29, 31, 33, 35, 37, and 39 Hz) using a Powerplate Pro5 (Netherlands) device. Each vibration session will last for 10 seconds, with a 5-second rest interval between frequencies.
* The Achilles tendon will be percussed 10 times with an electronic reflex hammer.

ELIGIBILITY:
Inclusion Criteria:

* DXA T-scores ≤-2.5 (osteoporotic) or T-scores > -1 (no bone loss)
* Individuals who agree to participate in the study

Exclusion Criteria:

* History of musculoskeletal surgery within the past year
* Individuals with health conditions that severely affect mobility
* Vestibular disorders
* Visual impairments
* Other rheumatic, psychiatric, or severe neurological diseases
* Chronic decompensated cardiac, renal, or hepatic insufficiency
* Panic attacks
* Individuals with skin lesions on the soleus muscle
* History of fractures or prostheses in the lower extremities
* History of kidney stones
* 2+ or more edema in the lower extremities, lymphedema
* History of malignancy
* History of osteomalacia or vitamin D deficiency

Ages: 60 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Bone myoregulation reflex latency | Through study completion, an average of 8 weeks.
  The measurement will be taken as the time difference between the moment of mechanical stimulation and the onset of the reflex response in the EMG. The unit of measurement for latency is milliseconds.
Bereitschafts (Readiness) Potential | Through study completion, an average of 8 weeks.
  It refers to the myoelectric activity in the tibialis anterior and soleus muscles just before jumping. The onset time of this myoelectric activity will be evaluated in milliseconds, and the amplitude of this activity will be measured in millivolts.

SECONDARY OUTCOMES:
Soleus H-reflex | Through study completion, an average of 8 weeks
  The soleus T-reflex elicited by percussing the Achilles tendon with an electronic reflex hammer will be recorded using EMG. The unit of measurement for latency is milliseconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Therapy Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Kalaoglu E, Faruk Bucak O, Kokce M, Ozkan M, Cetin M, Atasoy M, Ayture L, Karacan I. High-frequency whole-body vibration activates tonic vibration reflex. Turk J Phys Med Rehabil. 2023 Jan 11;69(1):46-51. doi: 10.5606/tftrd.2023.10854. eCollection 2023 Mar. PMID 37201009
- [Background] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Background] Kilic A, Soyturk G, Karaoglu A, Topkara Arslan B, Karacan I, Turker KS. A reliability study on the cumulative averaging method for estimating effective stimulus time in vibration studies. J Electromyogr Kinesiol. 2023 Jun;70:102768. doi: 10.1016/j.jelekin.2023.102768. Epub 2023 Mar 20. PMID 36965288
- [Background] Karacan I, Cakar HI, Sebik O, Yilmaz G, Cidem M, Kara S, Turker KS. A new method to determine reflex latency induced by high rate stimulation of the nervous system. Front Hum Neurosci. 2014 Jul 18;8:536. doi: 10.3389/fnhum.2014.00536. eCollection 2014. PMID 25100978
- [Background] Karacan I, Turker KS. Exploring neuronal mechanisms of osteosarcopenia in older adults. J Physiol. 2026 Jan;604(2):672-688. doi: 10.1113/JP285666. Epub 2024 Aug 9. PMID 39119811
- [Background] Kanis JA. Assessment of fracture risk and its application to screening for postmenopausal osteoporosis: synopsis of a WHO report. WHO Study Group. Osteoporos Int. 1994 Nov;4(6):368-81. doi: 10.1007/BF01622200. PMID 7696835